CLINICAL TRIAL: NCT04792749
Title: Clinical Effects of Metformin on Fertility-sparing Treatment for Early Endometrial Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong-Won Lee, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MetforminEndometrialCancer
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Endometrial Cancer Stage I
Keywords: Endometrial cancer; Metformin; Progestin; Fertility-sparing treatment
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin treatment (Experimental): Patients who receive metformin in addition to progestin therapy
  Interventions: Drug: Metformin
- Conventional treatment (No Intervention): Patients who receive progestin therapy only

INTERVENTIONS:
Drug: Metformin — Patients are given 750, 1500, and 2000 mgs of metformin per os daily (dose increases weekly, then maintain at 2000 mgs) in addition to 500 mgs of medroxyprogesterone acetate per os daily and levonorgestrel-releasing intrauterine device for the treatment of early stage endometrial cancer.
  Arms: Metformin treatment

SUMMARY:
The purpose of the study is to investigate the effects of metformin in addition to the conventional progestin therapy in the fertility-sparing treatment of early stage endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial cancer radiologic International Federation of Obstetrics and Gynecology (FIGO) stage IA patients
* Endometrioid endometrial cancer patients
* FIGO cellular differentiation grade 1 patients
* Patients who wish to preserve fertility
* Patients who understand that the recommended treatment of endometrial cancer is surgical treatment even in early stages, but still wish to preserve fertility and avoid surgical treatment
* Patients who have good performance status (Eastern Cooperation Oncology Group (ECOG) performance score equal to or greater than 3)
* Patients who are not contraindicated to the progestin therapy
* Patients who are not contraindicated to the use of metformin

Exclusion Criteria:

* Patients who have already received chemotherapeutic or radiotherapeutic treatments for endometrial cancer
* Patients whose disease is already advanced and not indicated for fertility-sparing treatment
* Patients whose tumor cellular differentiation grade is greater than FIGO grade 1

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment response rates | 3 months after the initiation of the treatment
  Measurements of the primary lesion by the RECIST criteria
Treatment response rates | 6 months after the initiation of the treatment
  Measurements of the primary lesion by the RECIST criteria
Treatment response rates | 9 months after the initiation of the treatment
  Measurements of the primary lesion by the RECIST criteria
Treatment response rates | 12 months after the initiation of the treatment
  Measurements of the primary lesion by the RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Won Lee, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No